CLINICAL TRIAL: NCT03822858
Title: Autologous, Bone Marrow-Derived Mesenchymal Stem Cell-Derived Neural Progenitor Cells (MSC-NP), Expanded Ex Vivo; Administered Intrathecally
Brief Title: Expanded Access to Intrathecal Administration of Autologous Mesenchymal Stem Cell-derived Neural Progenitors (MSC-NP) in Progressive Multiple Sclerosis
Status: Available | Type: Expanded Access
Sponsor: Tisch Multiple Sclerosis Research Center of New York (Other)
Responsible Party: Sponsor
Other Study IDs: TISCHMS-MSCNP-003
Record Dates: First submitted 2019-01-24; First posted 2019-01-30 (Actual); Last update posted 2025-08-17 (Actual); Status verified 2025-08

CONDITIONS: Multiple Sclerosis
Keywords: Mesenchymal Stem Cells; Neural Progenitors; Autologous; Bone Marrow; Multiple Sclerosis
MeSH Terms: conditions — Multiple Sclerosis

STUDY DESIGN:
Expanded Access Types: Treatment

INTERVENTIONS:
Drug: Intrathecal MSC-NP injection — Between 5 to 10 million MSC-NPs will be administered intrathecally in each dose.
  10 million cells is the maximum dose. Treatment will consist of 3-5 doses spaced 3 months apart.

SUMMARY:
To give expanded access to intrathecal autologous MSC-NP treatment to patients with progressive MS who do not meet the inclusion/exclusion criteria of our Phase II stem cell trial.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of MS as defined by the McDonald criteria
* Diagnosis of primary progressive or secondary progressive MS
* Patients will be 18 years or older
* Significant disability shown by an Expanded Disability Status Score (EDSS, [5]) ≥4.5 that was not acquired within the last 12 months *(Patients with moderate to severe cerebellar dysfunction who have an EDSS of <6.5 who are not eligible for our Ph II Version Date: 11/21/18 Version #4 9 study will be included. This is because EDSS scores are heavily related to muscle strength and not balance or coordination and most accurately reflect paraparesis. Also there are patients with MS who have disabling upper limb coordination dysfunction but EDSS scores of better than 6.5 who are not suitable for the Phase II study but may benefit from this therapy).
* Stable disease state as evidenced by a lack of gadolinium-enhancing lesions on an MRI and by a stable MRI disease burden (number of T2 lesions and size of lesions) in the last six months and no significant change in EDSS (1 point or more) in the last 12 months
* Does not qualify for the inclusion/exclusion criteria of our Phase II stem cell trial. For example, patients with EDSS >6.5 or MS symptom onset and/or duration of disease >15 years

Exclusion Criteria:

* All patients who have had any prior stem cell treatments, including HSCT
* Pregnant or nursing mothers or any woman intending to become pregnant in the next three years
* Use of systemic chemotherapeutic or anti-mitotic medications within three months of study start date due to the possibility of interference with bone marrow procedure
* History of central nervous system infection or immunodeficiency syndromes due to increased risk of CNS infection
* Patients who are anticipated to have difficultly accessing the intrathecal space related to scoliosis, obesity, or any other relevant factors determined by the PI.
* Patients who have not tried available therapies for their progressive MS

Ages: 18 Years to 70 Years | Sex: All
Age Groups: Adult, Older Adult

CONTACTS AND LOCATIONS:
Overall Officials: Saud A Sadiq, MD, FAAN, Principal Investigator — Tisch MS Research Center of New York
Locations (1):
- Tisch MS Research Center of New York, New York, New York, United States

REFERENCES:
- [Background] Harris VK, Stark J, Vyshkina T, Blackshear L, Joo G, Stefanova V, Sara G, Sadiq SA. Phase I Trial of Intrathecal Mesenchymal Stem Cell-derived Neural Progenitors in Progressive Multiple Sclerosis. EBioMedicine. 2018 Mar;29:23-30. doi: 10.1016/j.ebiom.2018.02.002. Epub 2018 Feb 3. PMID 29449193